CLINICAL TRIAL: NCT02756936
Title: Open Label, Randomized, Single Dose, Two-way Crossover Bioequivalence Study of Daclatasvir From Daclatasvir Zeta 60 mg Film Coated Tablets (Zeta Pharm Pharmaceutical Industries, Egypt) and Clatazev 60 mg Tablets (Bristol-Myers Squibb Pharma, UK) in Healthy Human Volunteers Under Fasting Condition.
Brief Title: Bioequivalence Study of Daclatasvir From Daclatasvir Zeta 60 mg Film Coated Tablets (Zeta Pharm Pharmaceutical Industries, Egypt) and Clatazev 60 mg Tablets (Bristol-Myers Squibb Pharma, UK)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genuine Research Center, Egypt (Industry)
Collaborators: Zeta Pharma Pharmaceutical Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GRC/1/16/600
Record Dates: First submitted 2016-04-28; First posted 2016-04-29 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Healthy
MeSH Terms: interventions — daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A Test (Experimental): Test drug (Daclatasvir zeta)1 tablet contains 60 mg Daclatasvir
  Interventions: Drug: Daclatasvir Zeta
- B Reference (Active Comparator): Reference drug (Clatazev)) 1 tablet contains 60 mg Daclatasvir
  Interventions: Drug: Clatazev

INTERVENTIONS:
Drug: Daclatasvir Zeta — 1 tablet contains 60 mg Daclatasvir
  Other Names: Daklinza
  Arms: A Test
Drug: Clatazev — 1 tablet contains 60 mg Daclatasvir
  Other Names: Daklinza
  Arms: B Reference

SUMMARY:
An open label randomized, single dose, two-way crossover bioequivalence study to determine the bioequivalence of Daclatasvir from Daclatasvir zeta 60 mg F.C.T ( Zeta Pharm Pharmaceutical Industries, Egypt) versus Clatazev 60 mg F.C.T (Bristol-Myers Squibb Pharma, UK) in Healthy Human Volunteers Under Fasting Condition

DETAILED DESCRIPTION:
Primary Pharmacokinetic Parameters: Cmax, AUC0→t and AUC0→∞ Secondary Pharmacokinetic Parameters: Ke, tmax and t1/2e. ANOVA using 5% significance level for transformed (with the 90% confidence intervals) and untransformed data of Cmax, AUC0→t and AUC0→∞ and for untransformed data of Ke, tmax and t1/2e.

The confidence intervals of logarithmically transformed Test/Reference ratios for Cmax, AUC0→t and AUC0→∞ to be within 80.00-125.00%.

A comprehensive final report will be issued upon the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, age 18 to 55 years, inclusive.
2. Body weight within 15% of normal range according to the accepted normal values for body mass index (BMI).
3. Medical demographics without evidence of clinically significant deviation from normal medical condition.
4. Results of clinical laboratory test are within the normal range or with a deviation that is not considered clinically significant by principal investigator.
5. Subject does not have allergy to the drugs under investigation.

Exclusion Criteria:

1. Subjects with known allergy to the products tested.
2. Subjects whose values of BMI were outside the accepted normal ranges.
3. Female subjects who were pregnant, nursing or taking birth control pills.
4. Medical demographics with evidence of clinically significant deviation from normal medical condition.
5. Results of laboratory tests which are clinically significant.
6. Acute infection within one week preceding first study drug administration.
7. History of drug or alcohol abuse.
8. Subject does not agree not to take any prescription or non-prescription drugs within two weeks before first study drug administration and until the end of the study.
9. Subject is on a special diet (for example subject is vegetarian).
10. Subject does not agree not to consume any beverages or foods containing methyl-xanthenes e.g. caffeine (coffee, tea, cola, chocolate etc.) 48 hours prior to the study administration of either study period until donating the last sample in each respective period.
11. Subject does not agree not to consume any beverages or foods containing grapefruit 7 days prior to first study drug administration until the end of the study.
12. Subject has a history of severe diseases which have direct impact on the study.
13. Participation in a bioequivalence study or in a clinical study within the last 6 weeks before first study drug administration.
14. Subject intends to be hospitalized within 3 months after first study drug administration.
15. Subjects who, through completion of this study, would have donated more than 500 ml of blood in 7 days, or 750 ml of blood in 30 days, 1000 ml in 90 days, 1250 ml in 120 days, 1500 ml in 180 days, 2000 ml in 270 days, 2500 ml of blood in 1 year.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Maximal measured plasma concentration (Cmax) | Up to 72 hours post dose in each treatment period
  Serial blood samples for determination of study drug will be collected at 0.00, 0.50, 1.00, 1.25, 1.50, 1.75, 2.00, 2.25, 2.50, 3.00, 3.50, 4.00, 6.00, 8.00, 12.00, 16.00, 24.00, 48.00, 72.00 hrs

SECONDARY OUTCOMES:
Time of the maximum plasma concentration (Tmax) | Up to 72 hours post dose in each treatment period
  he amount of time that a drug is present at the maximum concentration in serum

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshafeey, Ph.D. Pharma, Study Director — Genuine Research Center
Locations (1):
- Genuine Research Center GRC, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chow SC, Wang H. On sample size calculation in bioequivalence trials. J Pharmacokinet Pharmacodyn. 2001 Apr;28(2):155-69. doi: 10.1023/a:1011503032353. PMID 11381568
- [Background] Diletti E, Hauschke D, Steinijans VW. Sample size determination for bioequivalence assessment by means of confidence intervals. Int J Clin Pharmacol Ther Toxicol. 1991 Jan;29(1):1-8. PMID 2004861
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848
- See also: International conference of Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use. ICH Harmonized Tripartite Guideline. Guidelines for Validation of Analytical Procedures: Methodology. November, 1996 — http://www.pharmaweb.net/pwmirror/pw9/ifpma/ICH1.html